CLINICAL TRIAL: NCT02121613
Title: PERMIXON® 160 mg Hard Capsule Versus Placebo in the Treatment of Symptomatic Lower Urinary Tract Symptoms Due to Benign Prostatic Hyperplasia
Brief Title: PERmixon® in LUTS Evaluation Study (PERLES)
Acronym: PERLES
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pierre Fabre Medicament (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P00048 GP 4 04; 2014-000222-38 (EudraCT Number)
Record Dates: First submitted 2014-04-18; First posted 2014-04-23 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-09

CONDITIONS: Benign Prostatic Hyperplasia (BPH)
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — saw palmetto extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Permixon® 160 mg & Placebo (Experimental)
  Interventions: Drug: Permixon® 160 mg; Drug: Placebo matching Permixon® 160 mg; Drug: Placebo matching Tamsulosine LP
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo matching Permixon® 160 mg; Drug: Placebo matching Tamsulosine LP
- Tamsulosine LP & Placebo (Other): Active control arm
  Interventions: Drug: Tamsulosine LP; Drug: Placebo matching Permixon® 160 mg; Drug: Placebo matching Tamsulosine LP

INTERVENTIONS:
Drug: Permixon® 160 mg — Oral administration - 160 mg twice daily.
  Arms: Permixon® 160 mg & Placebo
Drug: Tamsulosine LP — Oral administration - 0.4 mg daily.
  Arms: Tamsulosine LP & Placebo
Drug: Placebo matching Permixon® 160 mg — Oral administration - twice daily.
Drug: Placebo matching Tamsulosine LP — Oral administration - daily.

SUMMARY:
The aim of this study is to support the efficacy of Permixon 160 mg b.i.d. in treating subjects with symptomatic Benign Prostatic Hyperplasia (BPH), compared to placebo, using Tamsulosine LP 0.4 mg as a reference treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male subject
* Between 45 and 85 years old
* Subject with bothersome lower urinary tract symptoms (LUTS) due to BPH such as frequency (daytime or night time), urgency, sensation of incomplete voiding, delayed urination or weak stream
* Subject naive to any prior treatment for LUTS due to BPH
* Prostate enlargement at digital rectal examination (DRE) suggestive of BPH
* I-PSS > 12 at enrolment visit and at inclusion visit
* QoL I-PSS score ≥ 3 evaluated at enrolment visit and at inclusion visit

Exclusion Criteria:

* Urological history such as urethral stricture disease and/or bladder neck disease, active (at enrolment and/or inclusion or recurrent urinary tract infection, stone in bladder or urethra)
* Any neurologic or psychiatric disease/disorder interfering with detrusor or sphincter muscle
* Insulin-dependent diabetes mellitus and non-controlled non insulin-dependent diabetes mellitus
* Known severe renal insufficiency or creatinine clearance < 30 ml/mn
* Known liver insufficiency or clinically significant abnormal liver function tests
* History of, or concomitant, cardiac arrhythmia or angina pectoris
* Orthostatic hypotension at enrolment or inclusion visit
* Known hypersensitivity to one of the constituents of the study drugs
* Is participating in another clinical trial

Ages: 45 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 833 (Actual)
Dates: Start 2014-04; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
International Prostate Symptom Score (I-PSS score) change | Day 180
  I-PSS score change from baseline to D180

CONTACTS AND LOCATIONS:
Overall Officials: Karim Keddad, MD, Study Director — Pierre Fabre Medicament
Locations (58):
- Czechia (7):
  - Benešov
  - Litoměřice
  - Pilsen
  - Prague
  - Roudnice nad Labem
  - Sternberk
  - Ústí nad Labem
- France (12):
  - Angers
  - Créteil
  - Limoges
  - Lyon
  - Marseille
  - Montreuil-Juigné
  - Nice
  - Nieul-sur-Mer
  - Paris
  - Saint-Orens-de-Gameville
  - Seysses
  - Tiercé
- Germany (12):
  - Berlin
  - Hagenow
  - Halle
  - Hamburg
  - Herzogenaurach
  - Hettstedt
  - Leipzig
  - Markkleeberg
  - Michelstadt
  - Mülheim
  - Nuremberg
  - Regensburg
- Italy (15):
  - Bari
  - Catanzaro
  - Foggia
  - Messina
  - Milan
  - Napoli
  - Novara
  - Orbassano
  - Padua
  - Palermo
  - Pesaro
  - Pietra Ligure
  - Prato
  - Roma
  - Udine
- Spain (12):
  - Barcelona
  - Coslada
  - El Palmar Murcia
  - Figueres
  - Getafe
  - Madrid
  - Parla
  - Sabadell
  - Salamanca
  - San Sebastián de los Reyes
  - Seville
  - Utrera de la Encomienda